CLINICAL TRIAL: NCT04528641
Title: A Phase 1, Dosage-Escalation Study to Assess the Safety and Immunogenicity of a COVID-19 Vaccine GRAd-COV2 in Healthy Adults and Elderly Subjects
Brief Title: Phase I Study to Assess the Safety and Immunology of a COVID-19 Vaccine With GRAd-COV2 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ReiThera Srl (Industry)
Collaborators: Istituto Nazionale per le Malattie Infettive "Lazzaro Spallanzani" IRCCS (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: RT-CoV-2
Record Dates: First submitted 2020-08-19; First posted 2020-08-27 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Phase I, open-label, dose escalation, clinical trial to assess the safety and immunogenicity of the candidate GRAd-COV2 vaccine in 90 healthy volunteers aged 18-55 years and elderly volunteers aged 65-85 years. The vaccine will be administered intramuscularly once in time.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm 1 - Low dose (Experimental): Arm-1 Healthy adult volunteers aged 18-55y will receive IM single dose of 5e10vp. N=15
  Interventions: Biological: GRAd-COV2
- Arm 2 - Intermediate dose (Experimental): Arm-2 Healthy adult volunteers aged 18-55y will receive IM single dose of 1e11vp. N=15
  Interventions: Biological: GRAd-COV2
- Arm 3 - High dose (Experimental): Arm-3 Healthy adult volunteers aged 18-55y will receive IM single dose of 2e11vp. N=15
  Interventions: Biological: GRAd-COV2
- Arm 4 - Low dose (Experimental): Arm-4 Healthy elderly volunteers aged 65-85y will receive IM single dose of 5e10vp. N=16
  Interventions: Biological: GRAd-COV2
- Arm 5 - Intermediate dose (Experimental): Arm-5 Healthy elderly volunteers aged 65-85y will receive IM single dose of 1e11vp. N=15
  Interventions: Biological: GRAd-COV2
- Arm 6 - High dose (Experimental): Arm-6 Healthy elderly volunteers aged 65-85y will receive IM single dose of 2e11vp. N=15
  Interventions: Biological: GRAd-COV2

INTERVENTIONS:
Biological: GRAd-COV2 — Single intramuscular administration.

SUMMARY:
RT-CoV-2 is a Phase I, open-label, dose escalation multicenter clinical trial to assess safety and immunogenicity of the candidate Coronavirus disease (COVID-19) vaccine GRAd-COV2 in Italian healthy volunteers aged 18-55 years and 65-85 years inclusive. GRAd-COV2 is based on a novel replication defective Gorilla Adenovirus and encodes for SARS-COV-2 Spike protein.

DETAILED DESCRIPTION:
RT-CoV-2 is a Phase I, open-label, dose escalation multicenter clinical trial to assess safety and immunogenicity of the candidate Coronavirus disease (COVID-19) vaccine GRAd-COV2 in Italian healthy volunteers aged 18-55 years and 65-85 years inclusive. GRAd-COV2 is based on a novel replication defective Gorilla Adenovirus and encodes for SARS-COV-2 full length prefusion stabilized Spike protein. GRAd-COV2 is developed and manufactured by ReiThera Srl.

This study will evaluate a singular intramuscular administration of GRAd-COV2 at 3 dose levels: 5e10, 1e11, 2e11viral particles (vp). There will be 6 study arms for a total of 90 healthy volunteers, divided into 2 cohorts of age, 18-55y and 65-85y, respectively.

Participants will be followed up for 24 weeks after vaccination. Follow up includes safety and immunogenicity assessment. Follow up visits will occur at day2, then 1, 2, 4, 8, 12, 24 weeks after vaccination.

The primary objective is to evaluate the safety and reactogenicity of a single dose vaccination schedule of GRAd-COV2 across 3 dosages in healthy younger and older adults. The secondary objective is to evaluate humoral and cellular immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following criteria to be eligible to participate in this study:

1. Provides written informed consent prior to initiation of any study procedures.
2. Be able to understand and agrees to comply with planned study procedures and be available for all study visits.
3. Agrees to the collection of venous blood per protocol.
4. Confirms to have not donated blood three months before the study
5. Agrees to refrain from blood during the study and until the three months after the end of the study.
6. Body Mass Index 18-29 kg/m2, inclusive, at screening.
7. Premenopausal women must agree to use one acceptable primary form of contraception.
8. Premenopausal women must have a negative urine pregnancy test the day of vaccination and are routinely using - and willing to use up to six months from vaccine administration - an effective method of birth control resulting in a low failure rate (i.e., hormonal contraception, condoms in combination with a spermicidal cream, male partner sterilization-vasectomy or total sexual abstinence).
9. Oral temperature ≤37.0 degrees Celsius the day of the administration of the vaccine
10. Pulse no greater than 100 beats per minute.
11. Systolic blood pressure (BP) is 85 to 139 mmHg, inclusive the day of vaccination.
12. Should not show laboratory values outside the normal range which may have clinical significance even in absence of specific signs or symptoms.

Exclusion Criteria:

A subject who meets any of the following criteria will be excluded from participation in this study:

1. Positive serology for anti-HIV-Ab
2. Positive HbBsAg
3. Positive anti-HCV-Ab
4. Positive for SARS-CoV-2 (either anti-S-Ab or anti-N-Ab)
5. Acute illness, as determined by the site PI or appropriate sub-investigator, the day of vaccination.
6. Breastfeeding women
7. Autoimmune and hyper-inflammatory condition
8. History of atopy (or any IgE associated condition) who had required treatment over the last 6 months;
9. History of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to any previous licensed or unlicensed vaccines;
10. Assumption of any immunomodulatory medication over the last 4 months (including, but not limited to, systemic corticosteroids, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar or toxic drugs). The use of low dose topical, ophthalmic, inhaled, and intranasal steroid preparations will be permitted.
11. Presence of self-reported or medically documented significant medical condition
12. Presence of self-reported or medically documented significant psychiatric condition
13. Significant cardiovascular disease needing therapy or history of myocarditis or pericarditis or heart surgery. Patients in treatment with Sartans or ACE-Inhibitors and good response to therapy may be included.
14. Neurological or neurodevelopmental conditions (e.g., history of migraines in the past 5 years, epilepsy, stroke, seizures in the last 3 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis or transverse myelitis).
15. Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell and squamous cell carcinoma of the skin, which are allowed.
16. Primary or secondary immunodeficiency of any cause.
17. Participated in another investigational study involving vaccination of biologic compounds in the last 12 months.
18. Currently enrolled in or plans to participate in another clinical trial with an investigational agent that will be received during the study-reporting period.
19. Administration of immunoglobulins and/or any blood or blood products within the 4 months before the first vaccine administration or at any time during the study.
20. Has any significant disorder of coagulation.
21. Has any chronic liver disease, including fatty liver.
22. Has a history of alcohol abuse or other recreational drug use within 6 months before the first vaccine administration.
23. Has any abnormality or permanent body art (e.g., tattoo) that would interfere with the ability to observe local reactions at the injection site (deltoid region).
24. Received or plans to receive additional vaccination within 4 weeks before or after each vaccination.
25. Has been reported as a case (confirmed or probable) of COVID-19 from the regional health system
26. Has any clinical conditions that, in the opinion of the site PI or appropriate sub-investigator, precludes study participation, this includes any acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Lanini, Principal Investigator — Istituto Nazionale per le Malattie Infettive "Lazzaro Spallanzani" IRCCS
Locations (2):
- Italy (2):
  - INMI Spallanzani, Rome
  - Centro Ricerche Cliniche, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capone S, Raggioli A, Gentile M, Battella S, Lahm A, Sommella A, Contino AM, Urbanowicz RA, Scala R, Barra F, Leuzzi A, Lilli E, Miselli G, Noto A, Ferraiuolo M, Talotta F, Tsoleridis T, Castilletti C, Matusali G, Colavita F, Lapa D, Meschi S, Capobianchi M, Soriani M, Folgori A, Ball JK, Colloca S, Vitelli A. Immunogenicity of a new gorilla adenovirus vaccine candidate for COVID-19. Mol Ther. 2021 Aug 4;29(8):2412-2423. doi: 10.1016/j.ymthe.2021.04.022. Epub 2021 Apr 23. PMID 33895322

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: a total of 180 subjects were screened and 98 subjects were enrolled in the study. seven out of 98 enrolled subjects were not administered vaccine because of withdrawal by subjects (3 subjects) and because the protocol allowed Screening period 21 days passed (4 subjects). a total of 91 subjects were administered vaccine.
Groups:
- Arm 4 - Low Dose: Arm-4 Healthy elderly volunteers aged 65-85y will receive IM single dose of 5e10vp. N=15
  GRAd-COV2: Single intramuscular administration.
Period: Overall Study
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Started | 15 | 15 | 15 | 16 | 15 | 15
Completed | 15 | 15 | 15 | 15 | 15 | 14
Not Completed | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose | Total
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 0 | 0 | 0 | 45
  >=65 years | 0 | 0 | 0 | 16 | 15 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (9.1) | 37.0 (10.2) | 36.2 (11.1) | 69.5 (4.6) | 70.8 (5.6) | 70.0 (3.5) | 53.1 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 6 | 5 | 5 | 5 | 33
  Male | 8 | 10 | 9 | 11 | 10 | 10 | 58
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 15 | 14 | 15 | 16 | 15 | 15 | 90
Region of Enrollment [Number; unit: participants]
  Italy | 15 | 15 | 15 | 16 | 15 | 15 | 91
Demographic - weight [Mean (Standard Deviation); unit: kg] | 73.9 (12.172) | 69.7 (14.91) | 70.9 (13.49) | 73.61 (12.874) | 70.37 (10.181) | 70.9 (10.54) | 71.59 (12.224)
Demographic - Height [Mean (Standard Deviation); unit: cm] | 173.3 (9.82) | 171.9 (10.93) | 173.8 (10.21) | 169.0 (9.01) | 168.1 (11.30) | 169.7 (9.47) | 170.9 (10.12)
Demographic - BMI [Mean (Standard Deviation); unit: Kg/m^2] | 24.514 (2.5747) | 23.367 (3.0412) | 23.332 (2.7751) | 24.767 (3.0552) | 24.574 (2.5569) | 25.035 (2.2006) | 24.514 (2.5747)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Solicited Local AE Signs and Symptoms 7 Days Following the Vaccination
Description: Participants were monitored for 7 days post-vaccination and the occurrence of solicited local AE signs and symptoms were collected.
Time Frame: 7 days following the vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
Participants
  Injection site pain | 10 | 12 | 10 | 2 | 1 | 4
  Injection site erythema | 1 | 2 | 2 | 0 | 0 | 1
  Injection site swelling | 0 | 0 | 1 | 0 | 0 | 1
  Injection site Haematoma | 0 | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Occurrence of Solicited Systemic AE Signs and Symptoms 7 Days Following the Vaccination
Description: Participants were monitored for 7 days post-vaccination and the occurrence of solicited systemic AE signs and symptoms were collected.
Time Frame: 7 days following the vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
Participants
  Headache | 5 | 6 | 10 | 6 | 3 | 2
  Fatigue | 8 | 7 | 10 | 7 | 2 | 4
  Pyrexia | 3 | 4 | 11 | 4 | 4 | 4
  Myalgia | 1 | 5 | 4 | 5 | 1 | 5
  Chills | 1 | 1 | 6 | 4 | 4 | 6
  Nausea | 2 | 2 | 3 | 1 | 3 | 2
  Neutropeonia | 1 | 1 | 2 | 1 | 1 | 2
  Abdominal Pain | 1 | 4 | 0 | 0 | 0 | 0
  Diarrhoea | 1 | 3 | 0 | 0 | 1 | 0
  Arthralgia | 0 | 0 | 0 | 0 | 0 | 1
  Back Pain | 0 | 0 | 0 | 1 | 0 | 0
  Cough | 0 | 0 | 0 | 0 | 0 | 1
  Faeces Soft | 0 | 0 | 1 | 0 | 0 | 0
  Hot flush | 1 | 0 | 0 | 0 | 0 | 0
  Hyperkalaemia | 0 | 0 | 0 | 0 | 1 | 0
  Muscle injury | 0 | 0 | 0 | 0 | 1 | 0
  Muscle strain | 0 | 0 | 0 | 0 | 0 | 1
  Tooth fracture | 0 | 0 | 1 | 0 | 0 | 0
  Dyspnoea | 0 | 0 | 0 | 0 | 0 | 1
  Oropharyngeal pain | 0 | 1 | 0 | 0 | 0 | 0
  Ecchymosis | 0 | 1 | 0 | 0 | 0 | 0
  Tooth abscess | 0 | 0 | 0 | 1 | 0 | 0
  Chalazion | 0 | 0 | 0 | 0 | 0 | 1
  Lymphadenopathy | 1 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Occurrence of Unsolicited AE 28 Days Following the Vaccination
Description: Occurrence of unsolicited AEs: unsolicited AEs were collected using the patient Diary and reported as "Any AE" occurring 28 days following the vaccination.
Time Frame: 28 days following the vaccination
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 - Low Dose: Arm-1 Healthy adult volunteers aged 18-55y will receive IM single dose of 5e10vp. N=14
  GRAd-COV2: Single intramuscular administration.
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
Participants
  week 1 - any AE : Mild | 9 | 9 | 13 | 9 | 6 | 7
  week 1 - any AE : Moderate | 3 | 5 | 6 | 1 | 2 | 2
  week 1 - any AE : Severe | 0 | 0 | 0 | 1 | 0 | 1
  week 2 - any AE: mild | 5 | 5 | 0 | 5 | 1 | 0
  week 2 - any AE: moderate | 0 | 1 | 0 | 0 | 1 | 0
  week 2 - any AE: severe | 0 | 0 | 0 | 0 | 0 | 0
  week 3 - Any AE: mild | 4 | 3 | 0 | 3 | 1 | 0
  week 3 - any AE: moderate | 0 | 1 | 2 | 1 | 1 | 0
  week 3 - any AE: severe | 0 | 0 | 0 | 0 | 0 | 0
  week 4 - any AE: mild | 1 | 2 | 0 | 0 | 1 | 0
  week 4 - any AE: moderate | 0 | 0 | 1 | 0 | 0 | 0
  week 4 - any AE: severe | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Occurrence of Serious AE 24 Weeks Following the Vaccination
Description: Occurrence of any treatment - emergent serious AE and treatment - emergent SAE related to study drug was monitored during the study period (24 weeks following vaccination)
Time Frame: 24 weeks following the vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
Participants
  Any treatment-emergent SAE related to study drug | 0 | 0 | 0 | 0 | 0 | 0
  Any treatment-emergent SAE | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Change in Leucocytes From Baseline
Time Frame: baseline, Weeks 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: 10^9 leucocytes /L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
10^9 leucocytes /L
  week 1 | -0.033 (1.285) | -0.199 (1.3799) | -0.265 (0.5758) | -0.159 (0.7563) | -0.019 (0.4475) | 0.055 (0.6884)
  week 2 | 0.218 (1.354) | 0.091 (1.2248) | -0.099 (0.6808) | 0.158 (0.9098) | 0.329 (0.7771) | 0.190 (0.6531)
  week 4 | -0.230 (1.2881) | 0.472 (1.2324) | -0.286 (0.6787) | -0.261 (1.0477) | 0.186 (1.0368) | 0.186 (1.1456)
  week 8 | 0.154 (0.8825) | 0.094 (1.2006) | -0.029 (1.0882) | -0.013 (0.8416) | 0.080 (0.5862) | -0.087 (0.6728)
  week 12 | -0.045 (1.0228) | 0.409 (1.7620) | 0.133 (1.1654) | -0.060 (0.9897) | 0.357 (0.8966) | -0.175 (0.7302)
  week 24 | -0.695 (1.199) | -0.125 (1.0887) | -0.263 (0.8854) | -0.310 (1.0615) | 0.196 (0.7996) | 0.199 (0.8817)

6. Primary Outcome: Change in Basophils From Baseline
Time Frame: Weeks 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: 10^9 basophils/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
10^9 basophils/L
  week 1 | -0.002 (0.0094) | -0.002 (0.0147) | -0.010 (0.0169) | -0.001 (0.0141) | -0.009 (0.0113) | -0.001 (0.0162)
  week 2 | 0.001 (0.0122) | 0.007 (0.0129) | -0.002 (0.0142) | 0.004 (0.011) | 0.003 (0.0272) | 0.004 (0.0124)
  week 4 | -0.004 (0.0118) | 0.0 (0.0120) | -0.003 (0.150) | 0.001 (0.054) | -0.003 (0.0129) | 0.004 (0.0199)
  week 8 | -0.001 (0.0122) | 0.001 (0.0133) | -0.001 (0.0119) | -0.002 (0.0164) | -0.005 (0.0092) | 0.003 (0.0116)
  week 12 | 0.002 (0.0142) | 0.003 (0.0159) | 0.0 (0.0108) | 0.0 (0.0121) | 0.0 (0.0156) | 0.002 (0.0142)
  week 24 | -0.004 (0.0135) | 0.004 (0.0112) | -0.001 (0.0146) | -0.003 (0.0168) | -0.004 (0.0140) | -0.001 (0.0141)

7. Primary Outcome: Change in Eosinophils From Baseline
Time Frame: Weeks 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: 10^9 eosinophils /L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
10^9 eosinophils /L
  week 1 | 0.009 (0.0478) | -0.017 (0.0649) | -0.007 (0.0555) | 0.031 (0.0483) | 0.009 (0.0674) | 0.006 (0.0467)
  week 2 | 0.014 (0.0370) | 0.029 (0.0644) | 0.024 (0.0697) | 0.046 (0.0574) | 0.037 (0.0743) | 0.021 (0.0439)
  week 4 | -0.013 (0.0873) | -0.003 (0.0603) | -0.003 (0.0471) | -0.008 (0.0680) | 0.001 (0.0442) | 0.027 (0.0870)
  week 8 | -0.023 (0.0716) | -0.002 (0.1202) | -0.033 (0.0979) | 0.010 (0.0732) | 0.006 (0.0617) | 0.021 (0.0935)
  week 12 | -0.004 (0.0840) | -0.017 (0.077) | -0.013 (0.1085) | -0.001 (0.0804) | 0.007 (0.0707) | 0.02 (0.0728)
  week 24 | -0.051 (0.0907) | -0.013 (0.0807) | 0.008 (0.1239) | 0.012 (0.0914) | 0.015 (0.0635) | 0.018 (0.0477)

8. Primary Outcome: Change in Neutrophils From Baseline
Description: Change from baseline was calculated as the value at each week minus the value at the baseline.
Time Frame: Weeks 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: 10^9 Neutrophils /L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
10^9 Neutrophils /L
  week 1 | -0.241 (1.1183) | -0.105 (1.3346) | -0.296 (0.5781) | -0.391 (0.7397) | -0.147 (0.3939) | -0.092 (0.5560)
  week 2 | -0.115 (1.1387) | -0.254 (1.0089) | -0.313 (0.4109) | -0.014 (0.8032) | -0.015 (0.5966) | -0.044 (0.4523)
  week 4 | -0.273 (1.3001) | -0.417 (1.0814) | -0.273 (0.4670) | -0.208 (1.0731) | 0.116 (0.8245) | 0.011 (1.0820)
  week 8 | -0.131 (0.8082) | 0.008 (1.1261) | 0.097 (0.9320) | 0.054 (0.7545) | -0.025 (0.4139) | -0.148 (0.5358)
  week 12 | -0.159 (0.8592) | 0.458 (1.8931) | 0.153 (1.0128) | 0.027 (0.9118) | 0.165 (0.6483) | -0.180 (0.6024)
  week 24 | -0.376 (1.1492) | -0.141 (0.8632) | -0.151 (0.6475) | -0.378 (0.9802) | 0.073 (0.6629) | 0.147 (0.7146)

9. Primary Outcome: Change in Monocytes From Baseline
Time Frame: Weeks 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: 10^9 Monocytes /L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
10^9 Monocytes /L
  week 1 | -0.0040 (0.0733) | -0.0227 (0.11218) | -0.0353 (0.0689) | -0.0525 (0.0668) | 0.0100 (0.0860) | -0.0307 (0.0694)
  week 2 | 0.0733 (0.1011) | 0.0427 (0.1353) | 0.0227 (0.1109) | 0.0144 (0.0999) | 0.0520 (0.0844) | 0.0280 (0.0820)
  week 4 | -0.0220 (0.0668) | -0.0327 (0.1142) | -0.0287 (0.0666) | -0.0556 (0.0909) | 0.0400 (0.1110) | -0.0193 (0.0656)
  week 8 | 0.0073 (0.0612) | 0.0113 (0.1336) | -0.0380 (0.0927) | -0.0431 (0.0624) | 0.0253 (0.0801) | -0.0227 (0.0849)
  week 12 | -0.0004 (0.0797) | 0.0007 (0.1331) | -0.0240 (0.0662) | -0.0475 (0.0772) | 0.0453 (0.0856) | -0.0387 (0.0605)
  week 24 | -0.0427 (0.0707) | -0.0107 (0.1163) | -0.0233 (0.1271) | -0.0227 (0.0960) | 0.0493 (0.1127) | -0.0021 (0.0567)

10. Primary Outcome: Change in Lymphocytes From Baseline
Time Frame: Weeks 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: 10^9 Lymphocytes /L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
10^9 Lymphocytes /L
  week 1 | 0.209 (0.5808) | -0.060 (0.4455) | 0.077 (0.2050) | 0.179 (0.2565) | 0.115 (0.2064) | 0.179 (0.2516)
  week 2 | 0.247 (0.3868) | 0.257 (0.3913) | 0.169 (0.4038) | 0.109 (0.2490) | 0.249 (0.2813) | 0.184 (0.3094)
  week 4 | 0.077 (0.4069) | -0.023 (0.3568) | 0.013 (0.2528) | 0.010 (0.3045) | 0.03 (0.2146) | 0.103 (0.1823)
  week 8 | -0.012 (0.3490) | 0.063 (0.3991) | -0.058 (0.2627) | -0.039 (0.2856) | 0.077 (0.2252) | 0.062 (0.2502)
  week 12 | 0.115 (0.4083) | -0.045 (0.3655) | 0.015 (0.2884) | -0.046 (0.3200) | 0.135 (0.2941) | 0.031 (0.2214)
  week 24 | -0.219 (0.3293) | 0.027 (0.5038) | -0.097 (0.2514) | 0.072 (0.2427) | 0.064 (0.2607) | 0.049 (0.3324)

11. Primary Outcome: Change in Erythrocytes From Baseline
Time Frame: Weeks 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: 10^12 Erythrocytes /L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
10^12 Erythrocytes /L
  week 1 | -0.091 (0.1603) | -0.067 (0.2342) | -0.037 (0.1574) | -0.0158 (0.2014) | -0.066 (0.2763) | -0.074 (0.1644)
  week 2 | 0.001 (0.01757) | -0.093 (0.220) | -0.037 (0.2251) | -0.084 (0.1660) | -0.073 (0.2447) | -0.149 (0.0896)
  week 4 | -0.065 (0.2011) | -0.059 (0.2081) | -0.039 (0.2599) | -0.059 (0.2024) | -0.119 (0.2456) | -0.079 (0.1122)
  week 8 | 0.026 (0.2133) | 0.002 (0.2320) | 0.047 (0.3186) | -0.024 (0.2767) | -0.061 (0.3035) | -0.034 (0.1874)
  week 12 | 0.054 (0.1722) | -0.036 (0.3260) | 0.027 (0.3375) | -0.013 (0.2587) | -0.045 (0.2680) | -0.070 (0.1488)
  week 24 | 0.007 (0.2073) | -0.046 (0.2601) | 0.001 (0.2936) | 0.018 (0.2453) | -0.058 (0.2505) | -0.062 (0.1691)

12. Primary Outcome: Change in Hematocrit From Baseline
Time Frame: Weeks 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: percentage of Total
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
percentage of Total
  week 1 | -1.16 (1.446) | -0.50 (2.429) | -0.35 (1.280) | -1.81 (2.05) | -1.38 (2.155) | -0.59 (1.499)
  week 2 | -0.19 (1.552) | -0.49 (2.086) | -0.33 (1.991) | -0.52 (2.004) | -0.80 (2.267) | -1.47 (0.647)
  week 4 | -0.59 (1.492) | -0.41 (2.004) | 0.15 (2.091) | -0.41 (2.339) | -1.26 (2.160) | -0.78 (0.986)
  week 8 | 0.26 (1.950) | .047 (2.132) | 0.85 (2.857) | -0.04 (2.790) | -0.91 (2.775) | 0.05 (2.017)
  week 12 | 0.31 (1.594) | -0.32 (3.175) | 0.61 (2.312) | -0.13 (2.819) | -0.49 (2.511) | -0.59 (1.470)
  week 24 | 0.21 (1.758) | -0.29 (2.534) | 0.62 (2.020) | 0.32 (2.511) | -0.81 (2.255) | -0.79 (1.389)

13. Primary Outcome: Change in Platelets From Baseline
Time Frame: Weeks 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: 10^9 Platelets /L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
10^9 Platelets /L
  week 1 | 7.7 (19.56) | -0.1 (24.38) | 1.5 (27.38) | -3.2 (16.20) | -8.1 (12.15) | 2.3 (21.86)
  week 2 | 17.4 (25.92) | 10.5 (33.06) | 20.3 (24.62) | 4.6 (17.77) | 2.7 (16.23) | 6.5 (14.79)
  week 4 | 4.3 (22.90) | -0.2 (22.27) | 6.1 (24.28) | -0.1 (22.93) | -1.8 (17.76) | 6.2 (16.23)
  week 8 | 11.0 (22.90) | 8.2 (31.41) | 14.2 (23.86) | -3.8 (24.07) | 2.0 (14.11) | 9.4 (28.11)
  week 12 | 15.9 (31.26) | 6.0 (30.25) | 13.3 (27.51) | -7.1 (21.05) | -6.3 (16.19) | 0.1 (17.94)
  week 24 | 11.3 (30.27) | 11.3 (36.34) | 5.9 (18.30) | -2.7 (31.25) | 1.9 (19.30) | -4.4 (24.42)

14. Primary Outcome: Change in Hemoglobin From Baseline
Time Frame: Weeks 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
g/L
  week 1 | -3.6 (5.21) | -2.1 (6.31) | -2.3 (4.89) | -4.5 (5.70) | -1.7 (7.07) | -2.2 (4.44)
  week 2 | -0.8 (5.54) | -2.6 (6.33) | -2.8 (6.14) | -3.3 (5.51) | -2.1 (7.45) | -3.0 (3.25)
  week 4 | -2.3 (5.86) | -4.8 (6.05) | -5.8 (6.66) | -1.6 (6.55) | -1.9 (7.52) | 1.5 (5.01)
  week 8 | 3.5 (6.15) | -2.9 (6.61) | -0.9 (8.20) | 0.3 (7.84) | -1.6 (9.45) | 2.4 (4.87)
  week 12 | -2.0 (4.93) | -2.6 (8.94) | 0.1 (8.71) | 1.8 (8.07) | 0.6 (7.89) | 0.3 (5.74)
  week 24 | -0.8 (6.13) | -3.1 (7.55) | 0.1 (8.09) | 2.8 (6.97) | -0.2 (7.88) | -0.1 (5.45)

15. Primary Outcome: Change in Sodium From Baseline
Time Frame: week 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
mmol/L
  week 1 | -0.1 (1.33) | 0.6 (2.06) | 0.3 (2.29) | 0.3 (1.65) | 0.6 (1.92) | 1.8 (1.97)
  week 2 | 0.6 (1.72) | 0.4 (2.32) | 0.3 (1.79) | 0.3 (221) | -0.5 (1.85) | 1.5 (1.96)
  week 4 | 0.5 (1.36) | -1.6 (1.96) | 0.1 (1.39) | -1.1 (1.18) | 0.6 (1.92) | 0.8 (2.21)
  week 8 | 0.0 (1.56) | -0.5 (1.81) | -0.1 (2.03) | -0.7 (182) | 0.5 (2.07) | 0.3 (2.26)
  week 12 | -0.2 (1.37) | -0.9 (1.25) | 1.1 (2.31) | -0.8 (1.84) | -0.2 (2.11) | 1.8 (1.47)
  week 24 | 0.8 (1.86) | -0.3 (2.19) | 1.8 (2.01) | 0.1 (1.85) | 0.9 (1.85) | 2.1 (2.14)

16. Primary Outcome: Change in Potassium From Baseline
Time Frame: week 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
mmol/L
  week 1 | 0.125 (0.3070) | -0.007 (0.3696) | 0.189 (0.4025) | 0.036 (0.3269) | 0.239 (0.5699) | -0.158 (0.3481)
  week 2 | 0.057 (0.2369) | -0.037 (0.2778) | 0.064 (0.2900) | -0.049 (0.4433) | -0.137 (0.4979) | -0.089 (0.3626)
  week 4 | 0.036 (0.3004) | -0.195 (0.2952) | 0.113 (0.34446) | 0.023 (0.4688) | -0.023 (0.4196) | -0.227 (0.3090)
  week 8 | -0.028 (0.3874) | 0.045 (0.3680) | 0.241 (0.3395) | -0.008 (0.4328) | 0.271 (0.3383) | -0.209 (0.3582)
  week 12 | 0.040 (0.4153) | -0.205 (0.4556) | 0.217 (0.2773) | 0.072 (0.3896) | 0.089 (0.2322) | -0.110 (0.2961)
  week 24 | 0.061 (0.2474) | 0.161 (0.2367) | 0.324 (0.2924) | 0.023 (0.2988) | 0.253 (0.410) | -0.190 (0.3313)

17. Primary Outcome: Change in Alkaline Phosphatase From Baseline
Time Frame: week 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
U/L
  week 1 | 2.1 (7.52) | 0.7 (4.92) | -3.7 (6.52) | -4.9 (4.89) | -0.7 (6.76) | 0.9 (6.94)
  week 2 | 0.5 (7.06) | 2.0 (6.63) | -4.7 (6.43) | -1.8 (5.39) | -4.3 (5.61) | 0.3 (7.62)
  week 4 | 1.3 (9.62) | -0.4 (5.74) | 3.6 (7.52) | -2.4 (6.31) | -2.7 (6.60) | 3.2 (4.21)
  week 8 | 5.0 (6.31) | 2.5 (5.36) | 1.1 (6.35) | -2.4 (5.94) | 3.5 (6.24) | 4.1 (5.65)
  week 12 | 2.7 (11.92) | 3.2 (5.91) | 3.9 (7.81) | -1.1 (5.48) | -2.1 (10.02) | 0.1 (6.02)
  week 24 | 1.7 (8.17) | 5.3 (9.49) | 3.3 (9.50) | -1.7 (7.01) | 2.1 (11.48) | 2.3 (8.48)

18. Primary Outcome: Change in Alanine Aminotransferase From Baseline
Time Frame: week 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
U/L
  week 1 | 1.3 (6.69) | 2.3 (6.33) | -0.2 (2.91) | -1.8 (2.44) | 4.3 (20.30) | 0.2 (3.55)
  week 2 | 2.7 (16.39) | 2.0 (5.13) | 2.5 (5.25) | -1.1 (3.26) | 2.6 (3.98) | 0.9 (3.68)
  week 4 | 1.1 (10.91) | 2.9 (3.81) | 0.9 (6.65) | 0.9 (3.96) | 0.1 (3.84) | 0.7 (4.43)
  week 8 | 1.2 (12.13) | 4.1 (6.08) | 0.1 (5.46) | -1.4 (5.26) | 0.8 (7.02) | -0.1 (2.99)
  week 12 | 6.9 (12.59) | 4.9 (6.33) | 3.9 (9.84) | -0.5 (8.22) | 0.4 (3.76) | -1.1 (3.23)
  week 24 | -0.7 (11.81) | 1.2 (4.20) | 0.3 (10.26) | 10. (3.38) | -0.3 (6.31) | -0.9 (3.83)

19. Primary Outcome: Change in Aspartate Aminotransferase From Baseline
Time Frame: week 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
U/L
  week 1 | -1.60 (4.982) | 0.40 (4.768) | -0.40 (2.898) | -1.38 (4.530) | 3.93 (11.738) | -1.33 (2.380)
  week 2 | 9.07 (32.288) | 0.29 (3.106) | 2.27 (3.262) | -2.44 (5.151) | 0.07 (3.150) | -0.80 (3.649)
  week 4 | -0.13 (4.518) | 2.53 (3.067) | 0.87 (4.015) | 0.69 (4.191) | 1.47 (3.720) | -0.93 (3.240)
  week 8 | 1.07 (4.480) | 1.20 (5.735) | 1.13 (3.623) | -2.50 (4.487) | 1.13 (4.340) | -0.93 (3.411)
  week 12 | 2.73 (6.147) | 2.47 (4.533) | 2.20 (4.109) | .194 (4.106) | -0.20 (3.986) | 0.13 (3.739)
  week 24 | 0.33 (6.091) | 0.87 (2.774) | 0.07 (5.391) | -1.53 (4.357) | 4.27 (18.763) | -0.29 (3.384)

20. Primary Outcome: Change in Direct Bilirubin Form Baseline
Time Frame: week 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
umol/L
  week 1 | 0.1026 (0.9712) | -0.3420 (0.9950) | -0.2622 (1.5375) | -0.0214 (1.0992) | 0.2280 (0.8878) | 0.2280 (0.8419)
  week 2 | 0.4140 (0.8857) | 4.5942 (17.8620) | -0.1482 (1.1559) | -0.1603 (0.6767) | -0.0684 (0.05040) | -0.0570 (0.7129)
  week 4 | 0.1140 (0.7907) | 0.3762 (0.9053) | -0.1710 (1.6503) | -0.0107 (0.7835) | 0.0570 (0.7331) | -0.1254 (0.8802)
  week 8 | 0.6498 (0.8155) | 0.2394 (0.9362) | -0.1026 (1.8449) | 0.0962 (1.1945) | 0.0570 (0.8783) | 0.1140 (0.6452)
  week 12 | 0.4789 (1.4059) | 0.1938 (0.9209) | -0.3534 (1.3718) | -0.1603 (0.8365) | -0.6270 (0.7720) | -0.0228 (0.8547)
  week 24 | 0.0114 (0.8610) | 0.0689 (0.9883) | -0.1482 (2.1081) | 0.1254 (0.9531) | -0.0342 (1.2181) | 0.1710 (0.6938)

21. Primary Outcome: Change in Bilirubin From Baseline
Time Frame: week 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
umol/L
  week 1 | 0.3534 (3.7254) | -1.1970 (3.7725) | 0.1048 (5.4294) | 0.0641 (4.2155) | -0.0228 (3.5705) | 0.5586 (2.8697)
  week 2 | 1.1286 (3.4315) | -0.1938 (3.5435) | -0.1824 (4.4841) | -0.4275 (2.54871) | -0.7980 (1.7181) | -0.7069 (2.5436)
  week 4 | -0.7068 (3.0527) | 1.0146 (3.526) | -0.2736 (6.4174) | 0.1176 (2.9557) | -0.0456 (2.7064) | -0.6954 (2.9706)
  week 8 | 2.1546 (3.7037) | 0.2280 (3.2820) | 0.2052 (7.1427) | 0.0534 (3.9465) | -0.5244 (3.0702) | -0.3192 (1.9269)
  week 12 | 1.9038 (6.9092) | 0.3078 (3.7354) | -0.6954 (5.6701) | -1.1222 (2.5108) | -2.6220 (2.8960) | -0.3420 (3.1431)
  week 24 | -0.7524 (2.8223) | 0.05586 (3.9258) | 23.9286 (91.7547) | -0.0114 (3.4670) | -0.3078 (4.4235) | -0.1954 (2.9227)

22. Primary Outcome: Change in Albumin Form Baseline
Time Frame: week 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
g/L
  week 1 | -2.45 (2.989) | -0.65 (2.370) | -1.70 (2.6376) | -1.67 (2.775) | 0.03 (2.343) | -0.64 (2.346)
  week 2 | -0.01 (2.334) | -0.83 (3.253) | -1.37 (2.943) | -1.03 (1.1885) | -0.73 (2.504) | -1.61 (1.739)
  week 4 | 0.62 (3.150) | -159 (2.035) | -0.08 (2.486) | -1.00 (2.055) | -1.53 (2.707) | -0.87 (2.408)
  week 8 | -0.23 (2.666) | -2.07 (2.587) | 0.71 (2.619) | -1.47 (2.587) | -2.43 (2.880) | -0.45 (2.770)
  week 12 | -0.86 (2.442) | -1.68 (2.815) | -0.25 (2.167) | -0.64 (2.2143) | -0.93 (1.617) | -0.13 (1.848)
  week 24 | -0.62 (2.155) | -2.56 (2.201) | -1.59 (2.630) | -1.21 (2.811) | -0.07 (3.501) | 1.21 (2.598)

23. Primary Outcome: Change in Creatinine Form Baseline
Time Frame: week 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
umol/L
  week 1 | -0.6483 (5.2878) | -2.9467 (5.8701) | 1.4733 (3.9908) | -4.0333 (8.5827) | 1.2963 (9.553) | -0.5304 (7.3491)
  week 2 | 1.5323 (5.3404) | -2.1805 (4.9992) | 2.1216 (37176) | 0.3315 (7.9125) | 0.3536 (5.9657) | -1.3555 (6.7561)
  week 4 | -2.3575 (4.4284) | -4.2432 (4.7511) | 1.6501 (5.2284) | -2.4310 (8.9600) | -1.8959 (6.6394) | -1.7680 (5.9017)
  week 8 | 2.2116 (6.3904) | -0.3536 (5.6088) | 2.4163 (3.0889) | -3.228 (8.9278) | -1.5912 (4.6442) | -2.1216 (5.4779)
  week 12 | 0.5893 (6.8610) | -2.8288 (5.5929) | 1.1787 (3.2680) | -3.0940 (10.4097) | -4.4789 (6.7279) | -3.2413 (5.6175)
  week 24 | -4.9504 (5.6088) | -2.0037 (4.6112) | -0.11799 (5.382) | -4.2432 (9.2244) | -3.1824 (5.9751) | -1.6417 (7.1888)

24. Primary Outcome: Change in Lactate Dehydrogenase From Baseline
Time Frame: week 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
U/L
  week 1 | -3.5 (12.69) | 0.5 (20.00) | 6.5 (15.62) | -10.8 (17.09) | -2.6 (19.82) | 0.9 (14.11)
  week 2 | 8.4 (35.25) | 1.4 (21.89) | 7.3 (17.99) | -7.0 (20.64) | -10.9 (13.17) | -5.7 (16.18)
  week 4 | -3.0 (16.46) | -1.7 (18.67) | 5.1 (15.34) | 2.1 (12.37) | 1.3 (17.54) | -3.9 (19.78)
  week 8 | -4.3 (10.31) | -2.4 (16.82) | 14.2 (24.40) | -11.2 (17.86) | 3.7 (37.19) | -4.2 (17.31)
  week 12 | -9.1 (13.48) | -3.8 (20.23) | 1.3 (16.86) | -10.1 (17.55) | -8.9 (15.95) | -3.4 (23.85)
  week 24 | -9.4 (18.26) | -3.3 (20.58) | -2.1 (12.06) | -10.0 (19.42) | -3.1 (22.96) | 2.4 (25.13)

25. Primary Outcome: Change in Urea Nitrogen From Baseline
Time Frame: week 1,2,4,8,12, and 24
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 15
mmol/L
  week 1 | 0.0571 (1.9802) | 0.0524 (1.5732) | -0.5712 (2.7988) | 0.1428 (2.0927) | -0.4712 (1.5268) | -0.3237 (2.4570)
  week 2 | 0.2951 (1.9132) | 0.5284 (2.2289) | -0.9377 (3.3246) | -0.2365 (2.2977) | 0.7854 (1.2804) | -0.6378 (2.4125)
  week 4 | 0.1571 (2.2931) | -0.1856 (1.6149) | -0.1428 (2.3668) | -0.3570 (2.0358) | -0.6474 (1.8290) | -0.5807 (2.3925)
  week 8 | -0.4522 (2.0612) | -0.0286 (1.5584) | -0.0952 (2.322) | -0.0759 (2.3484) | -1.0900 (2.3572) | 0.3237 (2.1001)
  week 12 | -0.0143 (1.8835) | 0.1000 (2.1727) | -0.6045 (2.6703) | 0.3525 (2.3561) | -0.4667 (2.1063) | -0.6426 (1.9342)
  week 24 | -0.0619 (1.7148) | 0.2667 (2.8833) | -0.5331 (2.3939) | 0.5379 (2.3910) | -0.2999 (1.5902) | -0.1989 (2.9145)

26. Secondary Outcome: Number of Participants With Positive, Negative or Indeterminate Seroconversion for Anti-s Antibody
Description: To assess the cellular and humoral immune response to SARS-CoV2 elicited by the vaccine
  Immunogenicity Result: Seroconversion for Anti-S Antibody
  Interpretation: n. of subjects positive, negative or indeterminate at week 1, 2, 4, 8, 12, and 24 after vaccination.
Time Frame: week 1, 2, 4, 8, 12, and 24
Population: * One subject in arm-1 low dose (adult cohort) had an asymptomatic infection around the time of vaccination. This was discovered post hoc, and this subject was excluded from all Immunogenicity Analysis Set(IAS).
  * One subject in Arm-4 low dose (elderly cohort) had a suspicious non-specific reactivity to the tests and was excluded from the IAS.
  * Other specification: % = Calculated as nr. of subjects within category divided by nr. of subjects with non-missing observation at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 14 | 15 | 15 | 15 | 15 | 15
Participants
  week 1: positive | 0 | 0 | 0 | 0 | 0 | 0
  week 1: negative | 14 | 15 | 15 | 15 | 15 | 15
  week 1: indeterminate | 0 | 0 | 0 | 0 | 0 | 0
  week 2: positive | 8 | 7 | 8 | 4 | 5 | 5
  week 2: negative | 6 | 7 | 6 | 10 | 7 | 9
  week 2: indeterminate | 0 | 1 | 1 | 1 | 3 | 1
  week 4: positive | 13 | 14 | 13 | 14 | 14 | 14
  week 4: negative | 1 | 0 | 2 | 1 | 1 | 1
  week 4: indeterminate | 0 | 1 | 0 | 0 | 0 | 0
  week 8: number analyzed (Participants) | 14 | 15 | 14 | 15 | 15 | 15
  week 8: positive | 13 | 14 | 14 | 10 | 12 | 13
  week 8: negative | 1 | 1 | 0 | 3 | 3 | 1
  week 8: indeterminate | 0 | 0 | 0 | 2 | 0 | 1
  week 12: number analyzed (Participants) | 14 | 15 | 14 | 15 | 15 | 15
  week 12: positive | 13 | 13 | 13 | 10 | 11 | 13
  week 12: negative | 1 | 2 | 1 | 4 | 4 | 2
  week 12: indeterminate | 0 | 0 | 0 | 1 | 0 | 0
  week 24: number analyzed (Participants) | 14 | 13 | 13 | 12 | 13 | 13
  week 24: positive | 10 | 7 | 11 | 6 | 5 | 10
  week 24: negative | 4 | 4 | 1 | 6 | 6 | 3
  week 24: indeterminate | 0 | 2 | 1 | 0 | 2 | 0

27. Secondary Outcome: Number of Participants With Positive, Negative Anti-n Antibody
Description: To assess the cellular and humoral immune response to SARS-CoV2 elicited by the vaccine
  cellular and humoral immune parameters evaluated: anti-N Antibody Interpretation: n. of subjects positive, negative at week 1, 2, 4, 8, 12 and 24 compared to baseline
Time Frame: week 1, 2, 4, 8, 12 and 24
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 14 | 15 | 15 | 15 | 15 | 15
Participants
  week 1: positive | 0 | 0 | 0 | 0 | 0 | 0
  week 1: negative | 14 | 15 | 15 | 15 | 15 | 15
  week 2: positive | 0 | 0 | 0 | 0 | 0 | 0
  week 2: negative | 14 | 15 | 15 | 15 | 15 | 15
  week 4: positive | 0 | 0 | 0 | 0 | 0 | 0
  week 4: negative | 14 | 15 | 15 | 15 | 15 | 15
  week 8: positive | 0 | 0 | 0 | 0 | 0 | 0
  week 8: negative | 14 | 15 | 15 | 15 | 15 | 15
  week 12: number analyzed (Participants) | 14 | 15 | 14 | 15 | 15 | 15
  week 12: positive | 0 | 0 | 0 | 0 | 0 | 0
  week 12: negative | 14 | 15 | 14 | 15 | 15 | 15
  week 24: number analyzed (Participants) | 14 | 13 | 13 | 12 | 13 | 13
  week 24: positive | 0 | 0 | 0 | 0 | 0 | 0
  week 24: negative | 14 | 13 | 13 | 12 | 13 | 13

28. Secondary Outcome: Number of Participants With Positive, Negative for Micro Neutralization Test
Description: To assess the cellular and humoral immune response to SARS-CoV2 elicited by the vaccine cellular and humoral immune parameters evaluated: Micro Neutralization test
  Interpretation: n. of positive and negative subjects at week 4 and week 24 by evaluating geometric mean titer change from baseline
Time Frame: week 4 and week 24
Population: number of subjects analyzed is calculated based on number of subjects with non missing observation thus numbers of subjects analyzed may vary between the observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 14 | 15 | 15 | 15 | 15 | 15
Participants
  positive week 4 | 6 | 10 | 9 | 12 | 10 | 11
  Negative week 4 | 8 | 5 | 6 | 3 | 5 | 4
  Positive week 24: number analyzed (Participants) | 14 | 13 | 13 | 12 | 13 | 13
  Positive week 24 | 2 | 4 | 5 | 2 | 4 | 6
  Negative week 24: number analyzed (Participants) | 14 | 13 | 13 | 12 | 13 | 13
  Negative week 24 | 12 | 9 | 8 | 10 | 9 | 7

29. Secondary Outcome: Immunogenicity - T-cell Response
Description: To assess the cellular and humoral immune response to SARS-CoV2 elicited by the vaccine cellular and humoral immune parameters evaluated.
  T-cells were evaluated on frozen and fresh (week2) samples
  Within-cohort comparisons to assess the difference in immune response according to different doses in the same population Across-the-cohort comparison to assess whether elderlies and adults have a different pattern of immune response after vaccination at different endpoints
  Unit: spot-forming cells [SFC]/1 × 10^6 peripheral blood mononuclear cell [PBMC]
  Interpretation: values higher than at baseline are indicative of a persistent spike-specific memory T-cell establishment.
Time Frame: baseline, week 2, week 4, week 8, week 12, week 24
Population: as for outcome 28
Measure: Median (Inter-Quartile Range); unit: SFC/1x10^6 PBMC
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
Number analyzed (Participants) | 14 | 15 | 15 | 15 | 15 | 15
SFC/1x10^6 PBMC
  T-cell response baseline | 54 [23.0 to 88.0] | 88.0 [43.0 to 138.0] | 128.0 [65.0 to 213.0] | 320.0 [78.0 to 760.0] | 165.0 [128.0 to 565.0] | 425.0 [295.0 to 1050.0]
  T-cell response week 2 (fresh samples) | 1161.0 [438.0 to 2430.0] | 2857.0 [412.0 to 4702.0] | 2272.0 [1243.0 to 3568.0] | 1917.0 [1353.0 to 3613.0] | 2262.0 [1228.0 to 3942.0] | 3142.0 [1555.0 to 8265.0]
  T-cell response week 2 (frozen samples) | 1214.0 [465.0 to 1475.0] | 1095.0 [328.0 to 3083.0] | 905.0 [743.0 to 1465.0] | 1258.0 [975.0 to 2790.0] | 1363.0 [570.0 to 2285.0] | 1618.0 [1010.0 to 5785.0]
  T-cell response week 4 | 788.0 [425.0 to 1353.0] | 1120.0 [368.0 to 2193.0] | 1330.0 [573.0 to 2285.0] | 1153.0 [745.0 to 2188.0] | 1258.0 [395.0 to 2000.0] | 1645.0 [1183.0 to 4215.0]
  T-cell response week 8 | 720.0 [355.0 to 945.0] | 948.0 [329.0 to 1468.0] | 1172.0 [628.0 to 1570.0] | 898.0 [403.0 to 1273.0] | 888.0 [353.0 to 1920.0] | 2133.0 [945.0 to 3538.0]
  T-cell response week 12 | 570.0 [458.0 to 733.0] | 655.0 [368.0 to 1073.0] | 856.0 [570.0 to 1553.0] | 898.0 [435.0 to 1670.0] | 835.0 [358.0 to 1278.0] | 1435.0 [760.0 to 2943.0]
  T-cell response week 24: number analyzed (Participants) | 14 | 13 | 13 | 12 | 13 | 13
  T-cell response week 24 | 538.0 [243.0 to 693.0] | 500.0 [238.0 to 918.0] | 798.0 [220.0 to 968.0] | 740.5 [529.0 to 936.5] | 643.0 [468.0 to 823.0] | 1223.0 [823.0 to 1930.0]

ADVERSE EVENTS:
Time Frame: Adverse Event occurred during the study period from enrollment to week 24
Description: Adverse events summarized by system organ class (SOC) and preferred term (PT), with number and percentage of subjects as well as the total number of occurrences.
  Adverse event summaries were ordered in terms of decreasing frequency for SOC and PT within SOC in the Total group and then alphabetically for SOC and PT within SOC. Summaries were ordered in terms of decreasing frequency for PT in the Total group in summaries where SOC was not included.
Arm/Group | Arm 1 - Low Dose | Arm 2 - Intermediate Dose | Arm 3 - High Dose | Arm 4 - Low Dose | Arm 5 - Intermediate Dose | Arm 6 - High Dose
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/16 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/16 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 12/15 | 14/15 | 14/15 | 13/16 | 9/15 | 9/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Low Dose (N=15) | Arm 2 - Intermediate Dose (N=15) | Arm 3 - High Dose (N=15) | Arm 4 - Low Dose (N=16) | Arm 5 - Intermediate Dose (N=15) | Arm 6 - High Dose (N=15)
Fatigue (General disorders) | 9 (31) | 7 (35) | 10 (11) | 7 (13) | 3 (4) | 4 (4)
injection site pain (General disorders) | 10 (11) | 12 (14) | 10 (10) | 2 (3) | 1 (1) | 4 (4)
Pyrexia (General disorders) | 3 (5) | 4 (6) | 11 (15) | 5 (6) | 4 (11) | 4 (4)
Chills (General disorders) | 1 (1) | 2 (2) | 6 (6) | 4 (7) | 4 (4) | 6 (7)
Injection Site Erithema (General disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Injection Site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site hematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (11) | 8 (16) | 11 (15) | 7 (10) | 3 (4) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 4 (4) | 6 (12) | 1 (1) | 5 (5)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 4 (4) | 3 (3) | 1 (3) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Faeces Soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropoenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premenstrual Syndrome (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate Aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkaliemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results will be agreed between ReiThera SRL and Istituto Nazionale per le Malattie Infettive Lazzaro Spallanzani. If one of the parties is interested in proceeding with a scientific publication, it must give written and electronic communication to the other party. Any impediments to publication must be communicated electronically within 30 days. If a party deems it inappropriate to publish, it will try to provide written changes to the text that could allow its publication.

DOCUMENTS (2):
  • Study Protocol (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT04528641/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT04528641/SAP_001.pdf